CLINICAL TRIAL: NCT02512094
Title: Validity and Reliability of Thai Version of Barthel Index for Hip Fracture Patients
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 236/2557(EC3)
Record Dates: First submitted 2015-07-26; First posted 2015-07-30 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Hip Fracture; Femoral Neck Fracture; Intertrochanteric Fracture
Keywords: Barthel index; Hip fracture; Validity; Reliability
MeSH Terms: conditions — Hip Fractures; Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Since an increasing in population age, there was an increasing in geriatric patients. Most of elderly patients needed rehabilitation programs to regain their quality of life during their medical treatments. Barthel index is a functional measurement to evaluate rehabilitation improvement in chronically-ill patients and also used for evaluation of patient's self-care.

Barthel index had been translated into many languages and validated in many medical conditions such as spinal cord injury, congestive heart failure, pneumonia, etc. However, Barthel index had not been translated into Thai language and validated to use in hip fracture patients.

The purposes of this study were to translate the Barthel index into Thai language and to assess validity and reliability of Thai version Barthel index in hip fracture patients.

DETAILED DESCRIPTION:
Since an increasing in population age, there was an increasing in geriatric patients. Most of elderly patients needed rehabilitation programs to regain their quality of life during their medical treatments. Barthel index is a functional measurement to evaluate rehabilitation improvement in chronically-ill patients and also used for evaluation of patient's self-care. This index had initially developed to evaluate the self-care of stroke patients which comprised of 10 questions about their basic activity of daily living. Barthel index had been well-accepted and widely used. Barthel index had been translated into many languages and validated in many medical conditions such as spinal cord injury, congestive heart failure, pneumonia, etc. However, Barthel index had not been translated into Thai language and validated to use in hip fracture patients.

Hip fractures was usually occured in geriatric patients and there was a trend to increase every year. Most of the hip fractures were treated by surgical methods which needed postoperative rehabilitation programs to regain their functions. Less than half of the patients with hip fracture could regain their functions to preoperative level. Therefore, these patients needed a specific questionnaire to evaluate their functions. Barthel index is an uncomplicated questionnaire and can be used to evaluate treatment outcome of the patients.

The purposes of this study were to translate the Barthel index into Thai language and to assess validity and reliability of Thai version Barthel index in hip fracture patients.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 50 years old
* Hip fractures within 2 weeks since injury

Exclusion Criteria:

* incommunicable patients
* pathological fractures
* multiple fractures or multiple trauma
* postoperative complications which change postoperative rehabilitation protocols

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hip fractured patients
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aasis Unnanuntana, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Elderly Hip Fracture: Age at least 50 years old Hip fractures within 2 weeks since injury
Period: Overall Study
Arm/Group | Elderly Hip Fracture
Started | 53
Completed | 53
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Elderly Hip Fracture
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Score of the Barthel Index
Description: Score of the Barthel Index ranging from 0 to 100 were collected when 0 is the minimum (worst outcome) and 100 is the maximum (best outcome).
  Score was reported as mean score of the Barthel Index.
Time Frame: up to 1 month
Population: All patients were analyzed using descriptive statistics.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elderly Hip Fracture
Number analyzed (Participants) | 53
units on a scale | 43 (14.4)

ADVERSE EVENTS:
Arm/Group | Elderly Hip Fracture
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No